CLINICAL TRIAL: NCT05528588
Title: Efficacy of Furoscix in Heart Failure Patients With Diuretic Resistance
Brief Title: Furoscix in Heart Failure Patients With Diuretic Resistance
Acronym: RESISTANCE-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: scPharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Ambarish Pandey, ASSISTANT PROFESSOR - Internal Medicine (Cardiology), University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0768
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients will undergo stratified randomization based on BAN-ADHF score (0-11 vs. ≥ 12). Within each stratum, patients will be randomized in a 1:1 ratio (intervention: control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ≥ 12 BAN-ADHF, Furoscix (Experimental): Patients with diuretic resistance as determined by a BAN-ADHF score ≥ 12 will receive Furoscix over 5 hours at 8 mg/mL.
  Interventions: Combination Product: Furoscix
- <= 11 BAN-ADHF, Furoscix (Experimental): Patients without diuretic resistance as determined by BAN-ADHF score <= 11 will receive Furoscix over 5 hours at 8 mg/mL.
  Interventions: Combination Product: Furoscix
- ≥ 12 BAN-ADHF, control (Active Comparator): Patients with diuretic resistance as determined by a BAN-ADHF score ≥ 12 will receive home dose oral diuretic.
  Interventions: Drug: Diuretic Therapy
- <= 11 BAN-ADHF, control (Active Comparator): Patients without diuretic resistance as determined by BAN-ADHF score <= 11 will receive home dose oral diuretic
  Interventions: Drug: Diuretic Therapy

INTERVENTIONS:
Combination Product: Furoscix — Study Drug: Furoscix®, (Furosemide Injection), 80 mg/10 mL is a proprietary furosemide formulation that is buffered to a neutral pH to enable subcutaneous administration and contained in a prefilled Crystal Zenith® (CZ) cartridge.
  Study Device: The Infusor is a compact, ethylene oxide (EtO) sterilized, single-use, electro-mechanical (battery powered, micro-processor controlled), on-body subcutaneous delivery system based on the SmartDose® Gen II 10 mL (West Pharmaceutical Services).
  The Furoscix Infusor is an investigational drug-device combination product. The Infusor is applied to the abdomen via a medical grade adhesive and delivers a subcutaneous infusion of Furoscix through a pre-programmed, biphasic delivery profile with 30 mg (3.75 mL) administered over the first hour, followed by 12.5 mg (1.56 mL) per hour for the subsequent 4 hours (Total dose is 80 mg (10 mL) over 5 hours).
  Other Names: subcutaneous furosemide
  Arms: <= 11 BAN-ADHF, Furoscix; ≥ 12 BAN-ADHF, Furoscix
Drug: Diuretic Therapy — Patients will receive home dose oral furosemide or oral furosemide per standard of care.
  Arms: <= 11 BAN-ADHF, control; ≥ 12 BAN-ADHF, control

SUMMARY:
This will be a randomized, open-label pilot study of 70 patients with and without diuretic resistance who were recently admitted and discharged for acute decompensated heart failure with and oral diuretic regimen testing whether Furoscix is more effective at achieving post-discharge outpatient diuresis than standard of care. Diuretic resistance will be identified using the BAN-ADHF (BUN, creAtinine, NP-levels, Age, Diabetes and DBP, HF hospitalization, and atrial Fibrillation) score which has been integrated into the electronic health record. The score is integer-based with a score of ≥ 12 indicating diuretic resistance with high likelihood of poor outcomes. The primary outcome is diuretic efficacy as measured by volume of urine produced 8 hours after treatment and urine sodium levels (assessed hourly or per urination episode within 8 hours of treatment).

DETAILED DESCRIPTION:
Heart failure is one of the leading causes of hospitalization in the United States, contributing to over 1 million emergency department visits and nearly 1 million hospitalizations for HF annually. The estimated mean cost for HF was $11,552 in 2014, totaling an estimated $11 billion. Thus, strategies to reduce the burden of acute care use for patients with heart failure are necessary. Acute decompensation of heart failure is characterized by volume overload and is primarily treated with intravenous diuretics. However, inefficient and ineffective diuresis both during hospitalization and in the post-discharge environment predispose patients to frequent readmission and a worse prognosis. Importantly, there is heterogeneity in patient response to intravenous diuresis, with an estimated 20-50% of patients having poor response to initial IV diuretic therapy. Patients who are resistant to intravenous diuresis have increased risk of rehospitalization and mortality. Importantly, our group recently derived an integer-based risk score (BAN-ADHF score) to predict patients with low diuretic efficiency.

The investigators will screen eligible patients in the inpatient setting and schedule a research appointment within 14 days after discharge. At the research appointment, patients will be consented and undergo stratified randomization based on BAN-ADHF score (≥ 12 vs. <=11). Within each stratum, patients will be randomized in a 1:1 ratio (intervention: control). The intervention arm (Furoscix over 5 hours at 8mg/mL) will be compared to a usual care group (home oral diuretic dose prescribed by discharge physician). Patients will be monitored for 8 hours in the Clinical Research Unit post-drug administration for clinical safety and to measure clinical response. This study will take place at the Clinical Research Unit in the Aston Building at UT Southwestern Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients discharged after ward hospitalization for acute decompensated heart failure
* Able to be screened and enrolled within 14 days of hospitalization
* Recent echocardiogram (6 months or less)
* Discharged with home diuretic regimen

Exclusion Criteria:

* Chronic kidney disease stage 5 (eGFR<20) or End Stage Kidney Disease
* Systolic blood pressure <100
* ICU hospitalization within 3 months
* Inotrope use within last 3 months
* Home inotropes
* Electrolyte abnormalities on discharge
* Inadequate data for BAN-ADHF score
* Pregnant
* Prior heart transplantation or left ventricular assist device
* Low-output heart failure
* Concurrent use of non-loop diuretic
* Advanced liver disease
* Severe malnutrition
* Skin/Soft tissue condition precluding Furoscix
* Inability to collect urine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ambarish Pandey, MD, MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients who were recently hospitalized with ADHF within 14 days of their discharge who were prescribed diuretic therapy at discharge.
Pre-assignment Details: Enrollment was stratified by diuretic resistance based on the BAN-ADHF diuretic efficiency score with score ≥ 12 indicating diuretic resistance. The BAN-ADHF score was calculated using clinical parameters from the index admission.
Period: Overall Study
Arm/Group | ≥ 12 BAN-ADHF, Furoscix | <= 11 BAN-ADHF, Furoscix | ≥ 12 BAN-ADHF, Control | <= 11 BAN-ADHF, Control
Started | 23 | 12 | 23 | 12
Completed | 23 | 12 | 23 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oral Furosemide - With Diuretic Resistance: This group received oral furosemide and had diuretic resistance
- Oral Furosemide - Without Diuretic Resistance: This group received oral furosemide and was without diuretic resistance
- Subcutaneous Furosemide - With Diuretic Resistance: This group received subcutaneous furosemide and had diuretic resistance
- Subcutaneous Furosemide - Without Diuretic Resistance: This group received subcutaneous furosemide and was without diuretic resistance
- Total: Total of all reporting groups
Arm/Group | Oral Furosemide - With Diuretic Resistance | Oral Furosemide - Without Diuretic Resistance | Subcutaneous Furosemide - With Diuretic Resistance | Subcutaneous Furosemide - Without Diuretic Resistance | Total
Number analyzed (Participants) | 23 | 12 | 23 | 12 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (6.9) | 55.4 (6.6) | 57.5 (9.0) | 56.0 (8.4) | 57.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 4 | 19
  Male | 18 | 7 | 18 | 8 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 4 | 10
  Not Hispanic or Latino | 20 | 12 | 20 | 8 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BAN-ADHF Score [Median (Inter-Quartile Range); unit: units] — The BAN-ADHF score ranges from 0-26 (BAN-ADHF score: blood urea nitrogen, creatinine, natriuretic peptide levels, atrial fibrillation, diastolic blood pressure, hypertension and home diuretic, and heart failure hospitalization). Higher scores indicate greater diuretic resistance risk.
  units | 14 [12 to 15] | 6 [5 to 8.25] | 14 [13 to 15] | 8.5 [5.75 to 9.25] | 13 [9 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Post-treatment Urine Output as Measured by Cumulative Urine Output Within 1 Day.
Description: Post-treatment diuretic efficiency is measured by cumulative urine output in mL per mg of treatment, observed hourly through 8 hours following the administration of study therapy (Furoscix vs. oral furosemide).
Time Frame: 1 day
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/mg
Arm/Group | ≥ 12 BAN-ADHF, Furoscix | <= 11 BAN-ADHF, Furoscix | ≥ 12 BAN-ADHF, Control | <= 11 BAN-ADHF, Control
Number analyzed (Participants) | 23 | 12 | 23 | 12
mL/mg | 34.0 [29.0 to 38.9] | 29.8 [22.9 to 36.7] | 22.6 [17.6 to 27.6] | 30.1 [23.3 to 37.0]

2. Secondary Outcome: Post-treatment Peak Spot Urine Sodium Levels in 1 Day
Description: Post-treatment peak spot urine sodium levels assessed hourly over 8 hours post-treatment.
Time Frame: 1 day
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | ≥ 12 BAN-ADHF, Furoscix | <= 11 BAN-ADHF, Furoscix | ≥ 12 BAN-ADHF, Control | <= 11 BAN-ADHF, Control
Number analyzed (Participants) | 23 | 12 | 23 | 12
mmol/L | 100 [89 to 111] | 96 [80 to 112] | 83 [72 to 94] | 95 [79 to 112]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Safety endpoints included adverse clinical outcomes included 30-day emergency department (ED) visits or heart failure (HF) hospitalizations, and creatinine, estimated glomerular filtration rate, and hypo- or hyperkalaemia at the end of study visit.
Groups:
- Subcutaneous Furosemide: This arm received subcutaneous furosemide (n=35)
- Oral Furosemide: This group received oral furosemide.
Arm/Group | Subcutaneous Furosemide | Oral Furosemide
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 10/35 | 13/35
Other Adverse Events (participants affected / at risk) | 6/35 | 3/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Furosemide (N=35) | Oral Furosemide (N=35)
Emergency department visit or hospitalization for heart failure (Cardiac disorders) | 10 | 13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Furosemide (N=35) | Oral Furosemide (N=35)
Increase in creatinine > 0.3 from discharge to end-of-study visit blood test (Renal and urinary disorders) | 5 | 3
Potassium ≤ 3.0 (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT05528588/Prot_SAP_000.pdf